CLINICAL TRIAL: NCT03470259
Title: Detection of Thyroid Cancer and Central Lymph Node Metastases Using EMI-137 Enhanced Molecular Fluorescent Guided Imaging: a Multicentre Feasibility and
Brief Title: Precision Thyroid Cancer Surgery With Molecular Fluorescent Guided Imaging
Acronym: TARGET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL62817.042.17
Record Dates: First submitted 2018-02-21; First posted 2018-03-19 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Papillary Thyroid Cancer; Lymph Node Metastases
MeSH Terms: conditions — Thyroid Cancer, Papillary; Lymphatic Metastasis | interventions — Spectrum Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EMI-137 0.09mg/kg administration (Experimental): Three patients will be once administered with EMI-137 0.09 mg/kg. Thereafter the patient will be observed for an hour. Two hours after injection surgery will be performed and only ex-vivo imaging and spectroscopy will be performed of thyroid glands and lymph nodes with a multispectral Near Infrared Fluorescence (NIRF) camera system and spectroscopy system.
  After interim analysis will be decided if this dosage group has an adequate tumor-to-background ratio and dose extension will be performed.
  Interventions: Drug: IV adminstration of EMI-137; Device: Multispectral Fluorescence Reflectance Imaging; Device: Spectroscopy
- EMI-137 0.13mg/kg administration (Experimental): Three patients will be once administered with EMI-137 0.13 mg/kg. Thereafter the patient will be observed for an hour. Two hours after injection surgery will be performed and only ex-vivo imaging and spectroscopy will be performed of thyroid glands and lymph nodes with a multispectral Near Infrared Fluorescence (NIRF) camera system and spectroscopy system.
  After interim analysis will be decided if this dosage group has an adequate tumor-to-background ratio and dose extension will be performed.
  Interventions: Drug: IV adminstration of EMI-137; Device: Multispectral Fluorescence Reflectance Imaging; Device: Spectroscopy
- EMI-137 0.18mg/kg administration (Experimental): Three patients will be once administered with EMI-137 0.18 mg/kg. Thereafter the patient will be observed for an hour. Two hours after injection surgery will be performed and only ex-vivo imaging and spectroscopy will be performed of thyroid glands and lymph nodes with a multispectral Near Infrared Fluorescence (NIRF) camera system and spectroscopy system.
  After interim analysis will be decided if this dosage group has an adequate tumor-to-background ratio and dose extension will be performed.
  Interventions: Drug: IV adminstration of EMI-137; Device: Multispectral Fluorescence Reflectance Imaging; Device: Spectroscopy
- EMI-137 0.045mg/kg administration (Experimental): If we have a excellent tumor to background ratio ((tumor fluorescence)/(surrounding tissue fluorescence)) in the 0.09 mg/kg group, we will de-escalate back to a 0.045 mg/kg group to evaluate TBR and reduce possible tracer toxicity in a thyroid cancer population with 90% 20 year survival.
  Three patients will be once administered with EMI-137 0.045 mg/kg. Thereafter the patient will be observed for an hour. Two hours after injection surgery will be performed and only ex-vivo imaging and spectroscopy will be performed of thyroid glands and lymph nodes with a multispectral Near Infrared Fluorescence (NIRF) camera system and spectroscopy system.
  After interim analysis will be decided if this dosage group has an adequate tumor-to-background ratio and dose extension will be performed.
  Interventions: Drug: IV adminstration of EMI-137; Device: Multispectral Fluorescence Reflectance Imaging; Device: Spectroscopy

INTERVENTIONS:
Drug: IV adminstration of EMI-137 — Intravenous administration of the fluorescent tracer EMI-137 approximately two hours before incision. Thereafter will be an observational period of an hour.
  Other Names: IMP administration
Device: Multispectral Fluorescence Reflectance Imaging — A multispectral Near Infrared Fluorescence (NIRF) camera system sensitive for EMI-137 fluorescence will be used for only ex-vivo Multispectral Fluorescence Reflectance Imaging (MFRI) of the thyroid gland and/or lymph node compartment.
  Other Names: MFRI
Device: Spectroscopy — A spectroscopy system sensitive for EMI-137 fluorescence will be used for only ex-vivo spectroscopy of the thyroid gland and/or lymph node compartment.

SUMMARY:
Almost 50 % of papillary thyroid cancer (PTC) patients have central lymph node metastases (CLNM), which are associated with a high risk of persistent or recurrent disease. However, the practice of performing a prophylactic central lymph node dissection (PCLND) routinely remains controversial. The proponents argue that without a PCLND, PTC patients with positive lymph nodes have an increased risk of local recurrence, and postponed node dissection leads to with 5-6 fold higher risk of morbidity. If performed, PCLND in clinical node negative patients increases staging to pN1 in more than 50% of the cases without increasing survival. The complication rate in PCLND is lower when compared to a technically challenging re-exploration in recurrent disease, with reported incidences of 0.6% and 7.3-20%, respectively. Opponents of routine PCLND point out the lack of randomized clinical trials and object to treatment-induced hypo-parathyroidism and recurrent nerve damage for the N0 patients. Currently, no diagnostic tool is available which reliably identifies these patient categories. Therefore, there is a clear need for novel diagnostic imaging modalities that overcome this issue. Molecular Fluorescence Guided Surgery (MFGS) is potentially such a diagnostic tool. The administration of NIR fluorescent tracers can increase detection accuracy of cancer and nodal metastatic tissue using macroscopic MFGS. Therefore, we aimed to identify a GMP-produced near infrared (NIR) tracer that potentially has a high target-to-background ratio in PTC compared to normal thyroid tissue. Tyrosine-protein kinase Met (c-Met) is significantly upregulated at the protein level in PTC compared to normal thyroid tissue. The investigators therefore hypothesize that the GMP-produced NIR-fluorescent tracer EMI-137 (targeting c-Met, peak emission at 675 nm range) might be useful for intraoperative imaging of PTC and nodal metastases. The investigators' aim is to investigate if the administration of EMI-137 is a feasible approach to detect PTC nodal metastases. Ultimately, this method might be useful to improve patient selection for CLND. Eventually, we might also be able to visualize multifocality, more selective lateral neck dissections and asses residual tissue after thyroidectomy. Ultimately, all of these strategies may reduce overtreatment, morbidity, and costs while maintaining the same or better effectiveness with a lower recurrence rate and improved quality of life.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, eligible for surgery
2. Bethesda VI fine needle aspiration (FNA) thyroid or FNA proven PTC metastasis (primary or recurrence).
3. Scheduled to undergo central and/or lateral lymph node dissection with or without thyroidectomy as discussed in the Multi-Disciplinary Thyroid Board.
4. WHO performance score of 0-2.
5. Written informed consent.
6. Mentally competent person who is able and willing to comply with study procedures.
7. For female subjects who are of childbearing potential are premenopausal with intact reproductive organs or are less than two years post-menopausal:

   * A negative serum pregnancy test prior to receiving the tracer
   * Willing to ensure that she or her partner uses effective contraception during the trial and for 3 months thereafter.

Exclusion Criteria:

1. Pregnancy or breast feeding
2. Advanced stage thyroid cancer not suitable for surgical resection
3. Medical or psychiatric conditions that compromise the patient's ability to give informed consent
4. Concurrent anticancer therapy (chemotherapy, radiotherapy, vaccines, immunotherapy) delivered within the last three months prior to the start of the treatment
5. The subject has been included previously in this study or has been injected with another investigational medicinal product within the past six months
6. History of myocardial infarction (MI), TIA, CVA, pulmonary embolism, uncontrolled congestive heart failure (CHF), significant liver disease, unstable angina within 6 months prior to enrollment
7. Any significant change in their regular prescription or non-prescription medication between 14 days and 1 day prior to IMP administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The feasibility of Molecular Fluorescence Guided Surgery using EMI-137 | From tracer administration until after data analyses which will take up to 1.5year
  To determine the optimal dose of the c-Met targeting NIRF tracer EMI-137 for an adequate TBR in PTC lymph nodes metastases using 3, and possibly 4, different dosages op EMI-137.

SECONDARY OUTCOMES:
Safety of using EMI-137 through monitoring vital signs | 1 day
  To evaluate the safety of EMI-137 through monitoring vital signs for evaluating possible (severe) adverse events.
Safety of using EMI-137 through monitoring injection site | 1 day
  To evaluate the safety of EMI-137 through monitoring the injection site for evaluating possible (severe) adverse events.
Feasibility of MFGS for detecting nodal metastasis | Up to one year
  To evaluate the feasibility of MFGS for the assessment of PTC and nodal metastasis by calculating target-to-background ratio.
Feasibility of spectroscopy for detecting fluorescence of PTC and lymph nodes | Up to one year
  To determine the feasibility of ex vivo spectroscopy measurements of PTC and lymph nodes for quantification of the fluorescence signal of EMI-137
Validation of flourescence | Up to one year
  To correlate and validate fluorescence signals detected ex vivo with histopathology and immunohistochemistry by determining if high flourescence areas show tumorcells in pathological examination.
Distribution of EMI-137 | Up to 1.5 year
  To evaluate the distribution of EMI-137 on a microscopic level using fluorescence microscopy.
Sensitivity and specificity of EMI-137 | Up to 1.5 year
  To quantify sensitivity and specificity of EMI-137 for PTC and nodal metastasis in order to make a power size calculation for a possible subsequent diagnostic accuracy study.

CONTACTS AND LOCATIONS:
Overall Officials: Schelto Kruijfff, MD, PhD, Principal Investigator — University Medical Center Groningen; Gooitzen M van Dam, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metman MJH, Jonker PKC, Sondorp LHJ, van Hemel BM, Sywak MS, Gill AJ, Jansen L, van Diest PJ, van Ginhoven TM, Lowik CWGM, Nguyen AH, Robinson DJ, van Dam GM, Links TP, Coppes RP, Fehrmann RSN, Kruijff S. MET-receptor targeted fluorescent imaging and spectroscopy to detect multifocal papillary thyroid cancer. Eur J Nucl Med Mol Imaging. 2024 Jul;51(8):2384-2394. doi: 10.1007/s00259-023-06525-5. Epub 2023 Nov 29. PMID 38017325
- [Derived] Jonker PKC, Metman MJH, Sondorp LHJ, Sywak MS, Gill AJ, Jansen L, Links TP, van Diest PJ, van Ginhoven TM, Lowik CWGM, Nguyen AH, Coppes RP, Robinson DJ, van Dam GM, van Hemel BM, Fehrmann RSN, Kruijff S. Intraoperative MET-receptor targeted fluorescent imaging and spectroscopy for lymph node detection in papillary thyroid cancer: novel diagnostic tools for more selective central lymph node compartment dissection. Eur J Nucl Med Mol Imaging. 2022 Aug;49(10):3557-3570. doi: 10.1007/s00259-022-05763-3. Epub 2022 Apr 7. PMID 35389070